CLINICAL TRIAL: NCT06152068
Title: Insulin Resistance, Lipid Profile, CRP, IL-18 and Carotid Intima-Media Thickness (CIMT) Diameter in Obese Adolescents
Acronym: CIMT
Status: Completed | Type: Observational
Sponsor: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Andy Darma, MD, Principal Investigator and Medical Staf in Pediatric Gastroenterology, Universitas Airlangga
Other Study IDs: Forth ID
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Obesity, Adolescent
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity: Subjects with obesity were assessed with body mass index or BMI (calculated with body weight in kg divided by body height square in m). The subjects were determined to be obese if BMI value z-score > +2 SD of WHO child growth standard (assessed with WHO Anthroplus).
- non-obesity: Subjects non-obesity were assessed with body mass index or BMI (calculated with body weight in kg divided by body height square in m). The subjects were determined to be non-obesity if BMI value z-score < +2 SD of WHO child growth standard (assessed with WHO Anthroplus).

SUMMARY:
Carotid intima-media thickness (CIMT) is a marker for detecting endothelium dysfunction, and has become a non-invasive method that is very useful in detecting and evaluating subclinical atherosclerosis in obese children and adolescents. This method is very useful in visually detecting and monitoring changes in the intima and its medial thickness, and can also evaluate changes within the arterial wall in the absence of localized plaque. Previous research that was conducted found an increase in CIMT diameter in 44 of 59 obese adolescents. Obesity has a risk of increasing the diameter of CIMT which carries the risk of atherosclerosis. Obesity accompanied by insulin resistance, and metabolic syndrome has a greater risk of atherosclerosis. Currently, the prevalence of obesity in adolescents is increasing. Interleukin 18 is a group of interleukin 1 whose levels increase in chronic inflammatory processes such as obesity, metabolic syndrome, and type 2 diabetes mellitus. IL-18 levels increase in obesity with increased CIMT.

Assessment of cardiovascular risk in obese adolescents is still a challenge for health practitioners, to prevent cardiovascular complications in obese adolescents which can cause sudden death at a young age. It is necessary to assess changes in the cardiovascular system that can be identified early by knowing the CIMT diameter. However, there is no definite reference value so the CIMT can be used as a reference for the occurrence of subclinical atherosclerosis in obese adolescents. In the previous study, CIMT was not examined in non-obese adolescents, so the cut-off for CIMT in non-obese was not known. Therefore, we have the opportunity to research to determine the thickness of CIMT and determine the cut-off value of CIMT which is at risk of experiencing early atherosclerosis in the obese adolescent population.

DETAILED DESCRIPTION:
This research is a cross-sectional study with an analytical observational to examine Carotid Intima-Media Thickness (CIMT) in normal adolescents compared to obese adolescents. The research population was obese adolescents aged 13-18 years who study in Junior and Senior High School in Surabaya and Sidoarjo. The samples were research subjects, namely obese teenagers who met the inclusion criteria and exclusion criteria. The selection of research samples was carried out randomly. The number of research samples was based on previous research with adolescent subjects, obtaining a minimum sample size of 50.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (obese and normal)
* Aged 13-18 years old
* Not Smoking
* Not consumed alcohol and drugs

Exclusion Criteria:

* Suffering from infections, inflammation, autoimmune diseases, cancer, chronic diseases, and endocrine disorders
* consuming steroids or hormone therapy

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy adolescents
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Body weight | 5 months
  The data will be presented as mean +/- SD (standard deviation). The body weight will be measure with Seca electronic flat scale 813, in kg.
  (in grams) for subjects >24 months age.
Body height | 5 months
  The data will be presented as mean +/- SD (standard deviation). The body height was measured using stadiometer Seca 213 (in cm).
Body Mass Index (BMI) | 5 months
  BMI was calculated by dividing body weight (in kg) by body height square (in m) [body weight (kg)/body height2 (m2)], in kg/m2 unit. The data will be presented as mean +/- standard deviation (SD)
Blood pressure | 5 months
  blood pressure was measure using Omron Automatic Blood Pressure Monitor (Omron Health Care Co., Ltd, Japan) (in mmHg), by placing the cuff on the right arm, then pull and tighten it according to the size if the arm. After it was installed correctly (fasten and did not move), the power button on the digital tension tool was pressed, and then the microprocessor started to drive air pressure into the cuff, and then the value of blood pressures will appear in the manometer tube column. Systolic blood pressure measurement was performed in a sitting position after the subject had rested for 10 minutes. The data will be presented as mean +/- standard deviation (SD)
Fasting insulin | 5 months
  Blood samples were collected at 08.00-09.00 after the subject fasted for 12 hours through the median cubital vein. Ten ml of blood was taken. The blood sample collection was done by a laboratory's employers or a nurse who had been hired by the researchers. After the blood was taken, it was placed into a tube containing ethylenediaminetetraacetic acid (EDTA) for further analysis of Fasting insulin (FI). After that, the tube containing blood samples was placed in a cooling box for transport to the lab. The data will be presented as mean +/- SD, in μU/mL.

SECONDARY OUTCOMES:
Carotid Intima Media Thickness | 5 months
  A CIMT test uses ultrasound technology to create images of your artery layers.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Aisiyah Widjaja, Ph.D, Principal Investigator — Child Health Department, Faculty of Medicine, Universitas Airlangga
Locations (1):
- RS Bhayangkara Surabaya, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No